CLINICAL TRIAL: NCT04646096
Title: Multicenter Study for Robotic Arm-assisted THA 4.0 System with Integration of Pelvic Tilt and ROM Assessments: Implant Position Accuracy and the Hip Spine Relationship
Brief Title: Multicenter Study for Robotic Arm-assisted THA 4.0 System: Hip Spine Relationship
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: American Hip Institute (Other)
Collaborators: Stryker Orthopaedics (Industry); Hospital for Special Surgery, New York (Other)
Responsible Party: Principal Investigator, Benjamin Domb, MD, Medical Doctor, American Hip Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AHI-003
Record Dates: First submitted 2020-11-18; First posted 2020-11-27 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2025-01

CONDITIONS: Osteoarthritis, Hip; Hip Disease
Keywords: Robotic-assisted Total Hip Arthroplasty; MAKOplasty
MeSH Terms: conditions — Osteoarthritis, Hip

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Mako THA 4.0 group (Experimental): Hip system used: femoral stem (Accolade II), acetabular cup (Trident II or MDM if necessary), femoral head (ceramic or metal head compatible with Accolade II), acetabular insert (X3 Trident II or MDM liner when using MDM cup). Mako THA 4.0 software also will be used.
  Interventions: Device: MAKO THA 4.0 System

INTERVENTIONS:
Device: MAKO THA 4.0 System — Measure how the accuracy and precision of robotic arm-assisted total hip arthroplasty (THA) for placement accuracy of implant position in both the anterior and posterior approach.. The intervention will assess the precision of the MAKO system in placing hip components according to plan. It will compare hip angles executed by the Mako system intraoperatively with the 'gold standard' of 3D computer tomography (CT) scans.
  The postoperative CT scan can show the precision of the MAKO system by accurately determining the location of hip replacements in patients after surgery.

SUMMARY:
The current study is a multi-center study to assess precision and accuracy of the robotic system with new software.

DETAILED DESCRIPTION:
Robotic-arm assisted surgery aims to reduce errors and improve accuracy for implant position in total hip arthroplasty (THA). In THA implant positioning plays a pivotal role in good clinical outcomes and reduces long-term wear, therefore, technology has been developed to help surgeons achieve more accurate implant position consistently. Computer-assisted navigation provides surgeon with knowledge to help guide surgeons intra-operatively with some systems computed tomography (CT)-based, others fluoroscopy based, and others imageless systems. Computer navigation has been shown to accurately place components, but does not provide the ability for patient specific pre-operative planning that CT- based robotics allows. While some may argue that robotic-arm assisted THA is more accurate, others argue that the cost and learning curve associated with robotic-arm assisted THA is not more accurate with no long-term clinical benefits. Robotic arm-assisted THA has been shown to improve accuracy of component placement and reduce outliers. Kayani et al reviewed 100 cases performed by a single surgeon with 50 THAs performed manually and 50 robotic arm-assisted. In this study, Kayani did not find a learning curve associated with achieving accuracy using the robotic arm-assisted technology; however, there was a 12 case learning curve for both himself and his operating staff that increased operative time [9]. Nodzo et al evaluated the use of the robotic arm-assisted THA using post-operative CT scans and found that both the acetabular and femoral component position were significantly accurate when compared to the intra-op position. Kamara et al reviewed a single surgeon case series to assess acetabular accuracy and found that 76% of manual THAs were within the surgeons' target zone compared to 97% of his robotic arm-assisted THAs, concluding that adoption of robotic arm-assisted THA provided significant improvement in acetabular component positioning during THA. Similarly, Redmond et al found that although there was a learning curve associated with robotic arm-assisted THA, operative time decreased with experience and acetabular component outliers decreased suggesting that while there is a learning curve with robotic arm-assisted THA the clinical benefits are better implant positioning and decreased outliers. Illgen et al reported that the improved acetabular accuracy in robotic arm-assisted THA significantly reduced dislocation rates when compared to manual THA. Bukowski et al reported robotic arm-assisted THA clinical outcomes at a minimum of 1 year and found that patients who underwent a robotic arm-assisted THA has higher clinical outcomes compared to a manual group, however, there have been no large multicenter studies that assess clinical outcomes after robotic arm-assisted THA.

In conjunction with numerous other patient-specific and surgical factors, such as age, sex, comorbidities, surgical approach, component selection, and impingement, component positioning is often cited as an important factor in optimizing THA stability. Lewinnek et al. defined the "safe zone" for component position as 40⸰±10⸰ of cup inclination and 15⸰±10⸰ of cup anteversion to minimize dislocation risk. However, recent studies have shown that not only do components continue to dislocate when placed in this zone, but that the majority of THA dislocations are positioned in this safe zone to begin with. Compounding this issue is the growing body of evidence showing that the acetabular component is not static in nature, as was the assumption with Lewinnek's safe zone, but rather dynamically changing with movement of the pelvis and spine during postural and positional changes. Alterations of the dynamic relationship between the hip, spine, and pelvis in patients with hip-spine pathology during movements such as transitioning from standing to sitting affects typical pelvic biomechanical accommodation, resulting in THA component impingement, instability, and dislocation. Therefore, patients with spinopelvic pathology secondary to arthritis, spinal fusion, or spinal deformity are more prone to dislocation and revision following primary THA. The standard modality for assessing hip component position postoperatively is a 2D anteroposterior radiograph, due to low radiation dose and low cost. However, hip replacement components are placed in a 3-dimensional pelvis and femur, and therefore an anteroposterior radiograph alone may not give accurate information on the anteversion of the acetabular or femoral component. Studies have shown that cup anteversion measured with radiographs can have serious deviations with a substantial error range (mean deviation +1.74°, range -16.6° to 29.8°). This is attributed to the fact that radiographs cannot control for pelvic rotation and/or tilt. Recently a limited number of studies have started to use the other imaging modalities for understanding pelvic tilt in patients undergoing hip arthroplasty.

ELIGIBILITY:
Inclusion Criteria:

* Requires primary total hip arthroplasty surgery
* Willing and able to comply with postoperative follow up requirements
* at least 18 years of age
* sign an IRB approved informed consent

Exclusion Criteria:

* body mass index >40
* Skeletally immature
* patient with active infection or suspected latent infection in or about joint
* bone stock inadequate for support or fixation of the prosthesis
* Neuromuscular disorders, muscle atrophy, or vascular deficient in the affected limb
* Ankylosing spondylitis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2024-10-10 (Actual); Study Completion 2024-10-10 (Actual)

PRIMARY OUTCOMES:
Computed Tomography scan. Placement accuracy of acetabular cup and femoral stem | 6 weeks postoperatively
  Using computed tomography to assess placement accuracy, Measured in degrees

SECONDARY OUTCOMES:
Pelvic tilt | Preoperatively and postoperatively at 6 weeks and 1 year
  measured preoperatively and intraoperatively in sitting and standing positions
Virtual range-of-motion | Preoperatively and postoperatively at 6 weeks and 1 year
  measured preoperatively and intraoperatively in sitting and standing positions using virtual range of motion impingement modeling
Patient satisfaction | 1 year postoperative
  Measured in a scale of 0-10 to determine how satisfied a patient is with their procedure. A score of 10 indicates most satisfied, a score of 0 is least satisfied.
Harris Hip Score | preoperative and 1 year postoperative
  Questionnaire. A measure of functionality of the operated hip. Measured scale: 0-100. Lower score means worse functional outcome.
Forgotten Joint Score | 1 year postoperative
  Assess likelihood the patient has forgotten that they had a hip replacement. Measured scale: 0-100. Higher score means better feeling of normalcy.
Hip Disability and Osteoarthritis Outcome Score | 1 year postoperative
  Assess pain and function. Measured scale: 0-100. Higher the score, the greater the outcome and patient experience.

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin G Domb, MD, Principal Investigator — American Hip Institute
Locations (1):
- American Hip Institute, Des Plaines, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nodzo SR, Chang CC, Carroll KM, Barlow BT, Banks SA, Padgett DE, Mayman DJ, Jerabek SA. Intraoperative placement of total hip arthroplasty components with robotic-arm assisted technology correlates with postoperative implant position: a CT-based study. Bone Joint J. 2018 Oct;100-B(10):1303-1309. doi: 10.1302/0301-620X.100B10-BJJ-2018-0201.R1. PMID 30295538